CLINICAL TRIAL: NCT00901979
Title: A 12 Week Study in Patients With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLCQ908A2203
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (7):
- LCQ908 Dose 1 (Experimental)
  Interventions: Drug: LCQ908A; Drug: metformin
- LCQ908 Dose 2 (Experimental)
  Interventions: Drug: LCQ908A; Drug: metformin
- LCQ908 Dose 3 (Experimental)
  Interventions: Drug: LCQ908A; Drug: metformin
- LCQ908 Dose 4 (Experimental)
  Interventions: Drug: LCQ908A; Drug: metformin
- LCQ908 Dose 5 (Experimental)
  Interventions: Drug: LCQ908A; Drug: metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: metformin
- Sitagliptin (Active Comparator)
  Interventions: Drug: Sitagliptin; Drug: metformin

INTERVENTIONS:
Drug: LCQ908A
  Arms: LCQ908 Dose 1
Drug: LCQ908A
  Arms: LCQ908 Dose 2
Drug: LCQ908A
  Arms: LCQ908 Dose 3
Drug: LCQ908A
  Arms: LCQ908 Dose 4
Drug: LCQ908A
  Arms: LCQ908 Dose 5
Drug: Placebo
  Arms: Placebo
Drug: Sitagliptin
  Arms: Sitagliptin
Drug: metformin

SUMMARY:
This study will assess the effect of LCQ when added to metformin.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c from 7.0-10.0%, Stable Metformin dose

Exclusion Criteria:

* CHF Class III-IV, Liver disease

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 693 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Effect of LCQ on measures of glucose control | 12 weeks

SECONDARY OUTCOMES:
Changes in body weight and related measures | 12 weeks
Insulin sensitivity | 12 weeks
Safety and tolerability | 12 weeks

CONTACTS AND LOCATIONS:
Locations (67):
- United States (48):
  - Clinical Research Advantage, Mesa, Arizona
  - Mesa Family Medical Center/Clinical Research Advantage, Mesa, Arizona
  - Woodland International Reserach Group, LLC, Little Rock, Arkansas
  - Associated Pharmaceutical Research, Buena Park, California
  - John Muir Clinical Research, Concord, California
  - *Private Practice*, Pasadena, California
  - Apex Research of Riverside, Riverside, California
  - California Research Foundation, San Diego, California
  - CNRI-San Diego, LLC, San Diego, California
  - Orange County Research Center, Tustin, California
  - Diablo Clinical, Walnut Creek, California
  - Denver VA Medical Center, Denver, Colorado
  - Complete Family Care, Northglenn, Colorado
  - Research Center Phase I-IV of Florida, Corp., Miami, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Perimeter North Medical Research, Roswell, Georgia
  - MacNeal Center for Clinical Research, Berwyn, Illinois
  - Venture Resource Group, Overland Park, Kansas
  - Cotton-O'Neil Clinical Research Center Topeka KS United States, Topeka, Kansas
  - Graves Gilbert Clinic Bowling Green KY United States, Bowling Green, Kentucky
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - Centennial Medical Group, Elkridge, Maryland
  - International Research Center Towson MD United States, Towson, Maryland
  - Fallon Clinic Worcester MA United States, Worcester, Massachusetts
  - Southwestern Medical Clinic, Bridgman, Michigan
  - Clarkston Medical Group, Clarkston, Michigan
  - Michigan State University - Kalamazoo Ctr for Med Studies, Kalamazoo, Michigan
  - Mississippi Medical Research, LLC, Picayune, Mississippi
  - ClinVest Research, Springfield, Missouri
  - St. John's Clinic - Medical Research, Springfield, Missouri
  - Montana Medical Research, Missoula, Montana
  - Meera Dewan, P.C., Omaha, Nebraska
  - Libra Clinical Research Associates, Brick, New Jersey
  - Physicians Research Center, Toms River, New Jersey
  - Endwell Family Physician, Endwell, New York
  - *Private Practice* Staten Island, Staten Island, New York
  - Medical Frontiers LLC, Carlisle, Ohio
  - Radiant Research, Greer, South Carolina
  - Southwind Medical Specialists Memphis TN United States, Memphis, Tennessee
  - Dallas Diabetic and Endocrinology Research Center, Dallas, Texas
  - Radiant Research - North Dallas, Dallas, Texas
  - Accurate Clinical Research, Houston, Texas
  - Blalock Clinical Research, Houston, Texas
  - Texas Center for Drug Development, P.A., Houston, Texas
  - Ettrick Health Center, Ettrick, Virginia
  - McGuire Veterans Medical Center, Richmond, Virginia
  - Northwest Clinical Research, Bellevue, Washington
  - Providence Physicians Group, Monroe, Washington
- Canada (8):
  - Health Sciences Centre - Diabetes Research Group, Winnipeg, Manitoba
  - Rivergrove Medical Clinic, Winnipeg, Manitoba
  - Credit Valley Prof Bldg, Mississauga, Ontario
  - Hamilton Medical Research Group, Sherbrooke, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Institut de Recherches Cliniques, Montreal, Quebec
  - Clinique Médicale Millénia Santé, Québec, Quebec
  - CHUS - Hopital Fleurimont, Sherbrooke, Quebec
- Italy (7):
  - Azienda Ospedaliera-Ospedali Riuniti di Bergamo, Bergamo
  - Centro Studi sull'Invecchiamento CeSI-Univers.G.D'Annunzio, Chieti
  - A.O.Polo Universitario Luigi Sacco, Milan
  - Istituto Scientifico San Raffaele - IRCCS, Milan
  - Ospedale S.Giovanni di Dio, Olbia
  - Presidio Ospedaliero di Cisanello Università degli Studi, Pisa
  - Univ.Tor Vergata - AUSL ROMA B - Sede Territoriale, Roma
- Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Oława, Poland
- Puerto Rico (3):
  - Policlinica Dr. Luis Rodriguez Carrasquillo, Carolina
  - Endocrine Lipid Diabetes Research Institute Ponce PR United States, Ponce
  - Miguel Sosa-Padilla, M.D., San Juan